CLINICAL TRIAL: NCT05903326
Title: Dexmedetomidine as a Sole Premedication for BMT Placement in Children Undergoing Bilateral Myringotomy Tube Placement Surgery
Brief Title: Dexmedetomidine as a Sole Premedication for BMT Placement
Acronym: BMT
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: NemoursANES
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Effect of Drug; Complication of Treatment
Keywords: Myringotomy Tube placement; Sedation and analgesia; Emergence delirium
MeSH Terms: conditions — Agnosia; Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- traditional treatment group: patients receiving bilateral myringotomy tube placement with the use of midazolam and intraoperative ketorolac
- New standard of care: patients receiving bilateral myringotomy tube placement with the use of dexmedetomidine alone
  Interventions: Other: Dexmedetomidine

INTERVENTIONS:
Other: Dexmedetomidine — this was an observational study only based on a change of practice
  Groups: New standard of care

SUMMARY:
There is very little evidence or research documenting any single method of sedation/analgesia for myringotomy tube (BMT) placement as being more effective than others. This was a retrospective chart review conducted to determine if there were significant differences in efficacy of administered pre-operative Midazolam and Intraoperative IM Ketorolac (traditional) vs. pre-operative Dexmedetomidine alone for pain and emergence delirium management of children undergoing placement of BMTs. The current protocol was changed under the direction of anesthesia and team members who wanted to see what the outcomes of the new management plan were. The plan was a prospective chart review and for this project, 276 patient charts were reviewed, 154 patients received traditional anesthesia treatment and 122 received Precedex. Data analysis indicated that the patients who had received Dexmedetomidine had significantly higher FLACC scores (meaning better pain control) than those who received the traditional therapy. There was no difference in emergence delirium between the two groups.

DETAILED DESCRIPTION:
Bilateral myringotomy tube placement (BMT) is one of the most frequently performed pediatric ENT surgeries. Ensuring adequate analgesia and anxiolysis during the perioperative period is essential, as agitation in children can lead to emotional distress for children and parents and can lead to complications such as injury and post-traumatic stress disorders. Premedication is vital for anxiolysis, as it can facilitate anesthesia induction by reducing agitation, enhancing cooperation, and minimizing fear, anxiety, and physical resistance during critical perioperative events such as parental separation, venipuncture, or mask application.

Standard perioperative analgesia and anxiolytic protocols for BMT vary by institution. Since the procedure is often performed without intravenous access, non-parental routes of administration are frequently used for both preoperative anxiolytic control and intraoperative analgesia. The popular perioperative analgesia regimen consists of intramuscular ketorolac, preceded by nasal midazolam before surgery for anxiolytic control. Midazolam is widely used as a pre-anesthetic medication due to its ability to reduce anxiety and ease parental separation fears while minimizing delay in discharge. Dexmedetomidine (Dex), an alternative medication with sedative and analgesic properties, has gained attention for its potential use in pediatric anesthesiology both for premedication and perioperative analgesia.

This study explored the efficacy of using preoperative intranasal dexmedetomidine as the sole alternative for providing both anxiolysis and perioperative analgesia compared to standard treatment. We aim to evaluate the efficacy and safety of dexmedetomidine as a premedication agent in pediatric patients undergoing BMT, potentially streamlining anesthetic protocols and enhancing the overall experience for pediatric patients, families, and perioperative clinical teams.

ELIGIBILITY:
Inclusion Criteria:

* healthy children between the ages of 6 months and 5 years who have had bilateral myringotomy tube placement without any other surgical procedures.

Exclusion Criteria:

* children who present for BMT coupled with other procedures
* children with coagulation disorders
* children with allergies to ketorolac or dexmedetomidine,
* ASA physical status classification greater than 2,
* children with sensory processing disorders and/or autism spectrum disorders or other emotional/behavioral problems which may affect pain scores or responses,
* children who undergoing placement of Triune myringotomy tubes
* children with medical conditions who would be at risk related to anesthesia or the surgical procedures itself.

Ages: 6 Months to 5 Years | Sex: All
Age Groups: Child
Study Population: healthy children between the ages of 6 months and 5 years who are undergoing BMT without any other procedure and not meeting any of the above exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
efficacy for pain and emergence delirium | preoperative period
  use of dexmedetomidine alone in preoperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Alfred I duPont Hospital for Children, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No
Data included retrospective chart review, with patients de-identified and coded upon completion of record-keeping. Data will be shared in aggregate format.

REFERENCES:
- [Background] Lee SJ, Sung TY. Emergence agitation: current knowledge and unresolved questions. Korean J Anesthesiol. 2020 Dec;73(6):471-485. doi: 10.4097/kja.20097. Epub 2020 Mar 25. PMID 32209961
- [Background] Mahmoud M, Barbi E, Mason KP. Dexmedetomidine: What's New for Pediatrics? A Narrative Review. J Clin Med. 2020 Aug 24;9(9):2724. doi: 10.3390/jcm9092724. PMID 32846947
- [Background] Pappas AL, Fluder EM, Creech S, Hotaling A, Park A. Postoperative analgesia in children undergoing myringotomy and placement equalization tubes in ambulatory surgery. Anesth Analg. 2003 Jun;96(6):1621-1624. doi: 10.1213/01.ANE.0000064206.51296.1D. PMID 12760984
- [Result] Robinson H, Engelhardt T. Ambulatory anesthetic care in children undergoing myringotomy and tube placement: current perspectives. Local Reg Anesth. 2017 Apr 19;10:41-49. doi: 10.2147/LRA.S113591. eCollection 2017. PMID 28458577
- [Result] Dave NM. Premedication and Induction of Anaesthesia in paediatric patients. Indian J Anaesth. 2019 Sep;63(9):713-720. doi: 10.4103/ija.IJA_491_19. PMID 31571684
- [Result] Behrle N, Birisci E, Anderson J, Schroeder S, Dalabih A. Intranasal Dexmedetomidine as a Sedative for Pediatric Procedural Sedation. J Pediatr Pharmacol Ther. 2017 Jan-Feb;22(1):4-8. doi: 10.5863/1551-6776-22.1.4. PMID 28337075
- [Result] Dewhirst E, Fedel G, Raman V, Rice J, Barry N, Jatana KR, Elmaraghy C, Merz M, Tobias JD. Pain management following myringotomy and tube placement: intranasal dexmedetomidine versus intranasal fentanyl. Int J Pediatr Otorhinolaryngol. 2014 Jul;78(7):1090-4. doi: 10.1016/j.ijporl.2014.04.014. Epub 2014 Apr 16. PMID 24814231